CLINICAL TRIAL: NCT07213180
Title: RETROUVE : Study of the Return to Driving in People Who Have Suffered a Cerebrovascular Accident (CVA)
Brief Title: Study of the Return to Driving in People Who Have Suffered a Cerebrovascular Accident (CVA)
Acronym: RETROUVE
Status: Completed | Type: Observational
Sponsor: Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de Kerpape (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01602-41; KER-2022_01 (Other: CMRRF de Kerpape)
Record Dates: First submitted 2024-01-10; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2024-01

CONDITIONS: Post-stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The RETROUVE study will provide healthcare professionals, patients and their families informations on the rate of return to driving in people who have suffered a stroke, and will provide a better understanding of the various factors that explain this return. This bi-centric study is being conducted in 2 parts: a retrospective part involving an analysis of medical records, and a prospective part involving a telephone questionnaire.

The main aim of this study is to assess the rate of return to driving in patients who have suffered a stroke, following an assessment of their fitness to drive. It will also aim to study the factors that explain a return to driving in post-stroke patients.

DETAILED DESCRIPTION:
This study aims to evaluate the rate of return to driving among stroke patients who underwent a formal fitness-to-drive assessment at the Kerpape CMRRF or Henry Gabrielle Hospital in 2019. Stroke patients may experience impairments in motor, cognitive, and executive functions, which can affect their ability to drive safely. The assessment involves a multidisciplinary evaluation including medical examination (vision, hearing, motor coordination), neuropsychological assessment (executive functions, attention, processing speed), and an on-road or simulator-based driving evaluation conducted by a driving instructor and occupational therapist.

The study consists of two phases:

Retrospective Analysis: Medical records of patients who underwent the driving assessment in 2019 will be reviewed. Collected variables include demographic characteristics (age, gender, education level), clinical data (stroke type, severity, comorbidities, medications affecting alertness), and driving assessment outcomes (favorable, unfavorable, or favorable with restrictions). The analysis will compare patients who were judged fit to drive with those who were judged unfit, in order to identify factors associated with a favorable driving outcome. Statistical methods include Chi-square tests, Student's t-tests or Wilcoxon tests depending on data distribution, and logistic regression to identify influential clinical, demographic, and driving-related factors.

Telephone Follow-Up: Approximately three years after the initial assessment, participants will be contacted by telephone to complete a follow-up questionnaire. The questionnaire evaluates current driving practices, limitations, perceived difficulties, and strategies adopted since the stroke. Telephone interviews are conducted by research staff and last approximately one hour.

All participants identified through medical records are informed about the study and their non-objection is recorded in the medical file. Data collection and analyses will adhere to the intention-to-treat principle. Missing data will be included in analyses, and any additional exploratory analyses will be clearly documented in the final report.

The study provides insight into long-term driving outcomes after stroke, the adaptation strategies patients implement, and the demographic and clinical factors influencing successful resumption of driving.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years and ≤ 85
* Having suffered a stroke (ischaemic and/or haemorrhagic)
* Having completed a driving assessment in 2019 at one of the 2 centres participating in the study
* Have not objected to taking part in the study

Exclusion Criteria:

* Protected adults (guardianship)
* Insufficient command of the French language
* Deceased patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients who have undergone a driving driving assessment in 2019 at CMRRF de Kerpape or at Kerpape or Henry Gabrielle Hospital
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Rate of return to driving after stroke | From date of stroke to date of driving assessment in 2019, assessed retrospectively.
  Proportion of stroke patients assessed as fit to drive (favorable decision) by the multidisciplinary team and the registered physician, based on the 2019 driving assessments at Kerpape CMRRF or Henry Gabrielle Hospital.
Demographic factors associated with return to driving | From date of stroke to date of driving assessment in 2019, assessed retrospectively.
  Age, gender, and education level of stroke patients, analyzed according to the opinion of the multidisciplinary team and the registered physician (favorable, unfavorable, or favorable with restrictions).
Clinical factors associated with return to driving | From date of stroke to date of driving assessment in 2019, assessed retrospectively.
  Clinical characteristics of stroke patients (stroke type, lesion side and date, comorbidities) analyzed according to the opinion of the multidisciplinary team and the registered physician (favorable, unfavorable, or favorable with restrictions).

SECONDARY OUTCOMES:
Evaluate the maintenance of driving three years after a stroke and any changes in driving habits and/or practices, as well as driving habits and/or practices, as well as any new strategies brought about. | From end of 2019 assessment to date of telephone questionnaire in 2022, assessed prospectively.
  This questionnaire will be sent to patients to gather information on their driving habits, limitations, fears and driving strategies.
  The aim is not to focus on the problem of accidents in post-stroke patients. Rather, the aim is to find out whether they were able to maintain their driving activity despite the onset of a stroke, and to identify any driving difficulties they encountered. We also want to see whether they have changed their driving habits and/or implemented new strategies. The demographic and clinical information we obtain about them will also enable us to identify the most influential factors in the recovery process.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BONAVENTUR, Study Director — CMRRF de Kerpape
Locations (1):
- Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de Kerpape, Ploemeur, Brittany Region, France